CLINICAL TRIAL: NCT00922467
Title: Closed-loop Delivery of Propofol and Remifentanil: Sparing Effect of Esmolol
Brief Title: Influence of Esmolol on a Closed-Loop Anesthesia System
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of effectiveness
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008/47
Record Dates: First submitted 2009-06-02; First posted 2009-06-17 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — esmolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): patients will receive a closed-loop administration of propofol and remifentanil according to bispectral level and a placebo
  Interventions: Drug: NaCl 9/00
- Esmolol (Experimental): patients will receive a closed-loop administration of propofol and remifentanil according to bispectral level and esmolol
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: NaCl 9/00 — Same volume as in the esmolol group
  Arms: Placebo
Drug: Esmolol — 1 mg/kg administrated over 10 minutes followed by an infusion of 0,2 mg/kg/hr during all the anesthetic period
  Arms: Esmolol

SUMMARY:
Main objective is to evaluate the sparing effect of esmolol on the required doses of propofol and remifentanil

ELIGIBILITY:
Inclusion Criteria:

* male patients scheduled for a general anesthesia

Exclusion Criteria:

* age lower than 18 years
* allergy to propofol, or to soja or to peanuts, or to sufentanil, to remifentanil, or to morphine, or to a myorelaxant or to an excipient,
* any other history of anaphylactic reaction,
* hypersensibility to sufentanil, or to remifentanil, or to other derivate of fentanyl,
* hypersensibility to esmolol or to an excipient,
* history of central nervous system disease,
* patients receiving a psychotropic treatment or an agonist-antagonist opiate,
* hypovolemic patients,
* patients receiving a cardio-vascular treatment,
* patients with a pacemaker,
* expected bleeding more than 20% of the blood volume,
* simultaneous general and loco-regional anesthesia,
* patients suffering from asthma, COPD, trouble of the heart rhythm or conduction, cardiac insufficiency, cardiogenogenic shock, Prinzmetal syndrome, pheochromocytoma,
* patients with a heart rate less than 50/min and/or an arterial hypotension,
* neurosurgical act or any other which precludes an adequate positioning of the bispectral electrode.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
administered doses of propofol and of remifentanil during anesthesia | end of anesthesia

SECONDARY OUTCOMES:
delay before recovery | at the end of anesthesia
hemodynamic abnormalities requiring a treatment | end of anesthesia
postoperative morphine requirement | Third post-anesthetic hour
explicit memorisation | Second postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (1):
- Hôpital Foch, Suresnes, France